CLINICAL TRIAL: NCT03481361
Title: Obstructive Sleep Apnoea (OSA) in Patients With Type 1 Diabetes (T1D): A Cross-Sectional Study
Brief Title: Obstructive Sleep Apnoea in Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Heart of England NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG_16-154; 209532 (Other: Integrated Research Approval System (IRAS))
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes; Obstructive Sleep Apnoea
Keywords: Obstructive sleep apnoea (OSA); Type 1 diabetes (T1D); Type 2 diabetes (T2D); Insulin-Dependent Diabetes Mellitus (IDDM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood serum and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to assess the relationship between obstructive sleep apnoea (OSA) and cardiac autonomic neuropathy (CAN) in patients with T1D.

The secondary aims of this study are to assess: (1) the prevalence of OSA in patients with T1D; (2) the relationship between OSA and metabolic parameters (such as glycaemic control, blood pressure, lipids and weight) in patients with T1D; (3) the relationship between OSA and diabetes-related microvascular complications (retinopathy, nephropathy, peripheral neuropathy) in patients with T1D; and (4) the potential mechanisms for the relationship between OSA and diabetic-related complications if such a relationship is found.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) has been reported to be very common in patient with type 2 diabetes (T2D), and this relation is expected as both conditions share obesity as a common risk factor. Despite that several articles have stated that OSA is an independent risk factor for abnormal glucose metabolism, hypertension, and cardiovascular diseases.

In contrast, patients with type 1 diabetes (T1D) are leaner and younger than patients with T2D, so it was expected that OSA might be less common in patients with T1D. However, few studies have reported the prevalence of OSA in T1D with a range between 8 and 46%. The relationship between OSA and diabetes-related vascular disease is poorly explored in patients with T1D. This suggests a mechanism other than obesity may be responsible for OSA in patients with T1D. Therefore, the investigators hypothesized that (1) OSA is related to CAN rather than obesity in patients with T1D. (2) OSA is common in patients with T1D. (3) OSA is associated with worse metabolic profile and microvascular complications in T1D. (4) Oxidative and nitrosative stress are possible mechanisms relating OSA to T1D complication.

ELIGIBILITY:
Inclusion Criteria:

* T1DM patient aged 18 and above, who was diagnosed more than 4 years ago.
* Able to give informed consent.
* Has sufficient proficiency in English to verbally answer interview questions.

Exclusion Criteria:

* Past medical history of severe respiratory disorders including treated OSA.
* Patients using oxygen supplements.
* Patients with end-stage renal disease receiving dialysis.
* Pregnancy.
* Dementia.
* End stage diseases with life expectancy below 6 months.
* Patients with implantable devices
* Patients with known atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with type 1 diabetes attending secondary care diabetes clinics at Heart of England NHS Foundation Trust (HEFT) in Birmingham.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
The relationship between OSA and cardiac autonomic neuropathy (CAN) in patients with T1D. | Single time point measurement (20- 30 min)
  CAN will be assessed using heart rate variability (HRV) and spectral analysis. During this test blood pressure and electrocardiogram (ECG) and will be recorded while resting in a sitting down position and during certain manoeuvres that include deep breathing and Valsalva, and standing up. The Result of this outcome will be categorized into normal, borderline, or abnormal.
  This study is one visit only, and the total duration of the visit is 2-4 hours. The time frame below is the approximate time needed to collect each outcome data.

SECONDARY OUTCOMES:
The prevalence of obstructive sleep apnoea in patients with T1D. | Single time point measurement (over 8 hours) at participant residence
  Sleep apnoea will be assessed using portable multi-channel home-based sleep device.
The relationship between the presence of OSA and metabolic profile in patients with T1D. | Single time point measurement (15 min)
  This outcome will be assessed by comparing the routine assessment results for patients with OSA to patients without OSA.
The relationship between OSA and the presence of microvascular complications in T1D patients. | Single time point measurement (1-2 hours)
  Microvascular complications include diabetic neuropathy, diabetic nephropathy, and diabetic retinopathy.
The potential mechanisms for the relationship between OSA and diabetic-related complications | Single time point measurement (about 5 min)
  Will be assessed using serum and plasma blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Abd Tahrani, MD, Principal Investigator — NIHR Clinician Scientist at University of Birmingham
Locations (1):
- Birmingham Heartlands Hospital, Heart of England NHS Foundation Trust, Birmingham, United Kingdom

REFERENCES:
- [Background] Borel AL, Benhamou PY, Baguet JP, Halimi S, Levy P, Mallion JM, Pepin JL. High prevalence of obstructive sleep apnoea syndrome in a Type 1 diabetic adult population: a pilot study. Diabet Med. 2010 Nov;27(11):1328-9. doi: 10.1111/j.1464-5491.2010.03096.x. No abstract available. PMID 20950392
- [Background] Golbidi S, Badran M, Ayas N, Laher I. Cardiovascular consequences of sleep apnea. Lung. 2012 Apr;190(2):113-32. doi: 10.1007/s00408-011-9340-1. Epub 2011 Nov 3. PMID 22048845
- [Background] Manin G, Pons A, Baltzinger P, Moreau F, Iamandi C, Wilhelm JM, Lenoble P, Kessler L, Kessler R. Obstructive sleep apnoea in people with Type 1 diabetes: prevalence and association with micro- and macrovascular complications. Diabet Med. 2015 Jan;32(1):90-6. doi: 10.1111/dme.12582. Epub 2014 Sep 25. PMID 25186832
- [Background] Reutrakul S, Van Cauter E. Interactions between sleep, circadian function, and glucose metabolism: implications for risk and severity of diabetes. Ann N Y Acad Sci. 2014 Apr;1311:151-73. doi: 10.1111/nyas.12355. Epub 2014 Mar 14. PMID 24628249
- [Background] Schober AK, Neurath MF, Harsch IA. Prevalence of sleep apnoea in diabetic patients. Clin Respir J. 2011 Jul;5(3):165-72. doi: 10.1111/j.1752-699X.2010.00216.x. Epub 2010 Jun 30. PMID 21679352
- [Background] Tahrani AA. Obstructive sleep apnea in patients with diabetes: implications for clinical practice. Diabetes Management. 2015; 5(6):511-23. doi: 10.2217/dmt.15.34.